CLINICAL TRIAL: NCT02412800
Title: Risk Factors of Postoperative Acute Lung Injury Following Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201412036RINC
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Acute Lung Injury
Keywords: Extravascular lung water; Pulmonary vascualr permeability index; Liver transplantation
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute lung injury: Postoperative acute lung injury was diagnosed according to the latest 2012 Berlin definition of acute respiratory distress syndrome by the PaO2/FiO2< 300 and acute onset of bilateral infiltrates on the chest radiograph that were not fully explained by cardiac failure during postoperative day 1 to postoperative day 3.

SUMMARY:
Postoperative acute lung injury (ALI) during the first 72 hours after liver transplantation is not uncommon. Injury may occur because liver transplantation is often associated with prolonged operative time, large volumes of fluid administration and transfusion, as well as inflammatory responses related to ischemia-reperfusion injury. For more precise perioperative fluid and hemodynamic management, modern monitoring systems, such as the pulse contour cardiac output (PiCCO) system, have been devised and reported in recent years. The PiCCO system uses the thermodilution technique to determine the cardiac index (CI) and thoracic fluid indices such as the intrathoracic blood volume index (ITBVI), extravascular lung water index (EVLWI), and pulmonary vascular permeability index (PVPI), all of which may reflect pulmonary fluid and injury status. However, perioperative changes in thoracic fluid indices in liver transplantation and their associations with postoperative ALI are not yet clear. In this study, the investigators aimed to determine patterns of change in perioperative thoracic fluid indices and compare these changes in recipients who did or did not develop postoperative ALI. Furthermore, the investigators will also try to determine the potential risk factors following liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* End stage liver disease receiving liver transplantation in NTUH.
* Age: 6 months old to 75 years old

Exclusion Criteria:

* history of pulmonary resection,
* chronic respiratory insufficiency
* cardiac dysfunction
* failure of the surgery.

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Liver transplant recipients in NTUH, Taipei, Taiwan. From 2004-2014.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative acute lung injury | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kuang Cheng Chan, M.D., Principal Investigator — Natioanal Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan